CLINICAL TRIAL: NCT03917290
Title: A Sports Injury Prevention Program to Reduce Subsequent Injuries After Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-2680
Record Dates: First submitted 2019-04-04; First posted 2019-04-17 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Brain Concussion; Musculoskeletal Injury; Locomotion; Postural Balance
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: Upon clearance to Return to Play (RTP) after concussion, all participants will be randomized to either a Neuromuscular training (NMT) group or usual care (no sports injury prevention training). Those in the NMT group will complete training for 20-30 minutes, two times per week, beginning at RTP and continuing at this frequency until the end of the current athletic season.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Upon clearance to RTP after concussion, participants randomized to NMT will complete training for 20-30 minutes, two times per week, beginning at RTP and continuing at this frequency for 8 weeks.
  Interventions: Behavioral: Neuromuscular training
- Usual Care (No Intervention): Participants cleared to RTP in the usual care arm will return to sports and not undergo any intervention.

INTERVENTIONS:
Behavioral: Neuromuscular training — Training will be conducted with a research assistant under the supervision of Dr. Howell (PI), a certified athletic trainer, who will meet with participants either at the individual or small group level (3-4 participants maximum). Training will be done within the Children's Hospital Colorado network-of-care locations, dependent on the location of participants. Due to in-person restrictions that have resulted from COVID-19, participants may also complete the intervention via remote (virtual) training sessions.
  Arms: Intervention

SUMMARY:
The long-term goal of this research is to implement methods that healthcare providers can use across diverse clinical settings to (1) identify athletes at risk for (musculoskeletal) MSK injury when cleared to return to play (RTP) after a concussion and (2) develop practical ways to reduce MSK injury risk following concussion RTP. The rationale is that once post-concussion MSK injury risk factors are known and prevention strategies tested, concussion RTP protocols will evolve to include injury risk reduction programs.

DETAILED DESCRIPTION:
Aims:

i. To determine the effect of a sports injury prevention program on MSK injuries initiated at concussion RTP and continued throughout the subsequent athletic season.

ii. To examine the effect of a neuromuscular training (NMT) program on clinical and instrumented postural control measures before and after the intervention.

The proposed study will use an intervention-based paradigm to further understand MSK injury risk after concussion RTP and to identify potential methods to reduce this risk. Common Data Element (CDE) and instrumented postural control data will be linked to objectively classify the clinical and functional underpinnings of concussion recovery and subsequent MSK injury among those engaged in an injury prevention program compared to those who are not. These are important elements to investigate because: 1) few studies have explored the mechanisms for MSK injury incidence after concussion using a multimodal and objective approach and 2) no investigations have examined interventions to improve long-term concussion outcomes initiated at RTP.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be those diagnosed with a concussion, defined as a brain injury caused by a direct blow to the head, face, neck or elsewhere on the body, resulting in the rapid onset of impairment of neurological function and diagnosed by Children's Hospital Colorado sports medicine physicians.
* Being between 12-18 years of age
* The ability to complete initial testing within 14 days of the injury
* A post-concussion symptom scale (PCSS) score of greater than 9 at the time of enrollment.

Exclusion Criteria:

* Active lower extremity injury affecting balance
* Pre-existing neurological disorder (bipolar disorder, schizophrenia, etc.)
* Previous concussion sustained within the past year
* Prisoners, pregnant females, individuals with limited decision-making capacity
* Pre-existing learning disability
* Structural brain injury (confirmed with neuroimaging)
* A high velocity injury mechanism (e.g motor vehicle accident).
* Less than one month remaining in the current athletic season.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Injury rate | One year
  The number of injuries / the number of exposures to sports injury following return to play (RTP) after concussion

SECONDARY OUTCOMES:
Physical activity level | <14 days post-concussion, and once the treating physician clears the subject for RTP, and 8 weeks after the treating physician clear the subject for RTP.
  In order to assess the effect of physical activity level on incidence and timing of subsequent musculoskeletal (MSK) injuries, we will provide participants with heart-rate activity monitors, worn from the initial post-concussion visit until RTP.
Dual-task walking speed. | <14 days post-concussion, and once the treating physician clears the subject for return to play (RTP), and 8 weeks after the treating physician clear the subject for RTP.
  Measure of the the average walking speed of subjects during dual-task conditions (m/s).
Reaction time | <14 days post-concussion, and once the treating physician clears the subject for RTP, and 8 weeks after the treating physician clear the subject for RTP.
  We will use smartphone-based reaction time assessments (ms)
Post Concussion Symptom Inventory | <14 days post-concussion, and once the treating physician clears the subject for RTP, and 8 weeks after the treating physician clear the subject for RTP.
  Overall symptom severity, rated as a sum score from 0-122. A higher score indicates more severe symptoms, while a 0 indicates that the patient is not experiencing symptoms.
PROMIS Short Form Pediatric 25 | <14 days post-concussion, and once the treating physician clears the subject for RTP, and 8 weeks after the treating physician clear the subject for RTP.
  A brief generalized quality of life questionnaire. We will calculate the sub-scale scores for the domains of Mobility, Depressive Symptoms, Anxiety, Peer Relationships, and Pain Interference. Each sub-scale is calculated as a sum of 4 questions, rated from 0-4. Thus, each subscale is from 0-16, where a 16 indicates a greater presence of the domain being measured.
Tampa Scale of Kinesiophobia | <14 days post-concussion, and once the treating physician clears the subject for RTP, and 8 weeks after the treating physician clear the subject for RTP.
  A brief questionnaire about fear of movement and injury related to returning to sport. The subject answers 18 questions rated from 1 (strongly disagree) to 4 (strongly agree). There is a total sum score ranging form 18-72, where a higher score represents more fear of movement.
Tandem gait | <14 days post-concussion, and once the treating physician clears the subject for RTP, and 8 weeks after the treating physician clear the subject for RTP.
  A brief assessment of gait performance included in the SCAT5. The outcome measure is time to complete the test.

OTHER OUTCOMES:
Compliance with NMT program | Week 1, 2, 3, 4, 5, 6, 7, and 8 of the NMT training program.
  The athletic trainer administering the protocol will record patient compliance for all treatment sessions. Each session is rated as yes/no by the supervising athletic trainer, and a total percentage of all training sessions is calculated as the compliance score.

CONTACTS AND LOCATIONS:
Overall Officials: David R Howell, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Howell DR, Seehusen CN, Carry PM, Walker GA, Reinking SE, Wilson JC. An 8-Week Neuromuscular Training Program After Concussion Reduces 1-Year Subsequent Injury Risk: A Randomized Clinical Trial. Am J Sports Med. 2022 Mar;50(4):1120-1129. doi: 10.1177/03635465211069372. Epub 2022 Jan 21. PMID 35060759
- [Background] Howell DR, Seehusen CN, Walker GA, Reinking S, Wilson JC. Neuromuscular training after concussion to improve motor and psychosocial outcomes: A feasibility trial. Phys Ther Sport. 2021 Nov;52:132-139. doi: 10.1016/j.ptsp.2021.05.014. Epub 2021 Aug 28. PMID 34482050